CLINICAL TRIAL: NCT00422929
Title: Eustachian Tube Growth and Development: Anatomy/Function
Brief Title: Eustachian Tube Growth and Development
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Margaretha L. Casselbrant, Professor, Otolaryngology, University of Pittsburgh
Other Study IDs: #0605009; 5P50DC007667-06 (NIH)
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Otitis Media
Keywords: otitis media; ear; acute otitis; middle ear; Eustachian tube; recurrent acute otitis media; chronic otitis media with effusion; no significant history of otitis media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cells obtained from buccal brushing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chronic otitis media with effusion (OME): history of chronic effusion (3 months if both ears, 6 months if one ear, or 3 episodes of effusion each lasting for 2 months or longer)
- recurrent AOM: recurrent acute otitis media (3 episodes in 6 months or 4 episodes in 1 year)
- no OM: no history of significant otitis media (i.e., does not meet criteria for chronic OME or recurrent AOM)

SUMMARY:
This study is to measure over time (from 3 years until 13 years of age) Eustachian tube function (the way the Eustachian tube works) and facial growth in groups of children with two types of middle-ear disease and with little past middle-ear disease. These measures will be used to determine if facial growth is related to improved Eustachian tube function, to see if the better function explains why young children who have middle-ear disease outgrow it as they get older, and to determine if these measures are different for the children in the three groups defined by disease history.

DETAILED DESCRIPTION:
The existing literature documents an important role for the Eustachian tube (ET) in the pathogenesis and/or persistence of otitis media (OM). Cross-sectional studies report a lower prevalence of OM in older children, a better ET pressure-regulating function in older children and age-related differences in ET form, length and width, and the vector orientation of the paratubal musculature. These growth-related changes in ET structural relationships are demonstrably predictive of increasingly more efficient ET function (ETF) and, because the ET and paratubal musculature are intimately related to the cranial base, the vector orientation of the ET system can be reconstructed from osteological or radiographic data. Together, these observations suggest that measurable, age-related changes in ET-paratubal muscle vector relationships are reflected in more efficient ETF and, by consequence, a decreased OM risk. The overall goal of the proposed longitudinal study is to evaluate the validity of this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* 3 years of age
* History of middle ear disease must fit into one of the 3 categories of ear history
* With or without patent tympanostomy tubes at time of entry
* Generally good health

Exclusion Criteria:

* Cleft palate or other syndromes predisposing to otitis
* History of significant orthodontic treatment or plan for such
* Cholesteatoma or other past ear surgery other than tubes
* Unable to cooperate for testing

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric otolaryngology clinic
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
change in Eustachian tube function | 5 years
  Eustachian tube function is tested yearly from age 3 years through age 7 years

SECONDARY OUTCOMES:
change in craniofacial measures | 5 years
  cross-correlations of anthropometric variables obtained by facial measurements, with growth over 5 years

OTHER OUTCOMES:
change in cephalometric variables | 5 years
  measurements obtained on cephalometric x-rays
change in later Eustachian tube function | 11 years
  Eustachian tube function tested yearly through 13 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha Casselbrant, MD, PhD, Study Director — University of Pittsburgh
Locations (1):
- ENT Research Center, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Casselbrant ML, Mandel EM, Seroky JT, Swarts JD, Doyle WJ. A pilot study of the ability of the forced response test to discriminate between 3-year-old children with chronic otitis media with effusion or with recurrent acute otitis media. Acta Otolaryngol. 2011 Nov;131(11):1150-4. doi: 10.3109/00016489.2011.603137. Epub 2011 Aug 17. PMID 21846295
- [Result] Casselbrant ML, Swarts JD, Mandel EM, Doyle WJ. The Cephalic Index is not different among groups of children aged 36-48 months with chronic otitis media with effusion, recurrent acute otitis media and controls. Int J Pediatr Otorhinolaryngol. 2013 Mar;77(3):334-7. doi: 10.1016/j.ijporl.2012.11.002. Epub 2012 Dec 30. PMID 23280277
- [Result] Casselbrant ML, Mandel EM, Seroky JT, Swarts JD, Doyle WJ. The forced-response test does not discriminate ears with different otitis media expressions. Laryngoscope. 2014 Nov;124(11):2619-23. doi: 10.1002/lary.24647. Epub 2014 Aug 11. PMID 24550093
- [Result] Swarts JD, Casselbrant ML, Teixeira MS, Mandel EM, Richert BC, Banks JM, El-Wagaa J, Doyle WJ. Eustachian tube function in young children without a history of otitis media evaluated using a pressure chamber protocol. Acta Otolaryngol. 2014 Jun;134(6):579-87. doi: 10.3109/00016489.2014.882017. PMID 24828350
- [Result] Mandel EM, Casselbrant ML, Richert BC, Teixeira MS, Swarts JD, Doyle WJ. Eustachian Tube Function in 6-Year-Old Children with and without a History of Middle Ear Disease. Otolaryngol Head Neck Surg. 2016 Mar;154(3):502-7. doi: 10.1177/0194599815620149. Epub 2015 Dec 1. PMID 26626132
- [Result] Casselbrant ML, Mandel EM, Doyle WJ. Information on co-morbidities collected by history is useful for assigning Otitis Media risk to children. Int J Pediatr Otorhinolaryngol. 2016 Jun;85:136-40. doi: 10.1016/j.ijporl.2016.03.040. Epub 2016 Apr 11. PMID 27240512
- [Result] Gremba AP, Weinberg SM, Swarts JD, Casselbrant ML. Craniofacial shape in children with and without a positive otitis media history. Int J Pediatr Otorhinolaryngol. 2016 May;84:110-5. doi: 10.1016/j.ijporl.2016.02.029. Epub 2016 Mar 5. PMID 27063764